CLINICAL TRIAL: NCT05944172
Title: Thoughts Content in OCD: What Links Between Mind Wandering and Obsessions
Brief Title: Impact of Attention on Obsessive Thoughts Through THOUGHT
Acronym: THOUGHTS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220613
Record Dates: First submitted 2023-02-10; First posted 2023-07-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obsessive Compulsive Disorder OCD
Keywords: OCD; wandering; daydreaming
MeSH Terms: conditions — Compulsive Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Impact of attention on obsessive through the THOUGHT-scale (Troublesome Human Obsessions and Untargeted General Habitual Thoughts Scale): a description of the content of thoughts according to the level of attention demanded by the environment in patients with obsessive disorder compulsive disorder (OCD) and patients without OCD" Validation of THOUGHTS.

DETAILED DESCRIPTION:
We developed a scale (the THOUGHTS) dedicated to allow a subject to subjectively measure its level of mind wandering/daydreaming (and obsessions in case of OCD patients) during different everyday situations. This scale is developed for 15 years old or older students (high school, university). Indeed, common point in everyday life was easier to find in students than in workers where lifestyle can be very divergent according to the job type. Through this scale, we will first detect the situations the more associated with mind wandering/daydreaming in healthy subjects. To do that, we will first find the 50% and the 25% of the situations the most associated with mind wandering. This step will allow us to distinguish two types of situations: situations with high level of mind wandering/daydreaming vs. situations with low level of mind wandering/daydreaming. Then we will do the same analyses in OCD patients to see if situations of high level of mind wandering are the same in both groups. Finally, we will compare the level of obsessions in OCD patients in these two types of situations (linked with high vs. low mind wandering, as defined by healthy subject, OCD patients and both populations).

To make these analyses, we will recruit 40 young OCD people (still students) from only one center, all diagnosed through DSM-5 criteria by a same senior and experimented child and adolescent psychiatrist and 40 matched healthy subjects.

For OCD patients: all comorbidities will be allowed except those associated with hallucinations or delusions: schizophrenia or bipolar disorder will then not be allowed. Neurological disorders will not be allowed too. Y-BOCS or CY-BOCS will be get and analyzed to find if severity could influence our results.

Healthy controls: they will be recruited to be matched with the OCD patients. No psychiatric or neurologic disorder will be allowed. No psychotropic or neurologic treatment will be allowed.

Finally, in terms of statistics, we will use non parametric tests.

ELIGIBILITY:
Inclusion Criteria:

For pathological patients:

* Over the age of 15
* Suffering from OCD (obsessive compulsive disorder)
* All comorbidities are possible except schizophrenia, bipolarity and anorexia nervosa
* Consultant or admitted to Albert Chenevier Hospital

For patients who are not affected by the disease:

* Over 15 years of age
* Consulted or admitted to GH Henri Mondor

Exclusion Criteria:

For pathological patients:

* Refusal to participate by the patient (and/or legal representative in the case of minors)
* Presence of schizophrenia, bipolar or anorexia nervosa

For patients who are free of these conditions:

* Presence of psychiatric or neurological pathology
* Refusal to participate on the part of the patient (and/or on the part of the legal representative in the case of minors)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 40 OCD patients 40 matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the obsession level (as measured by the THOUGHTS-scale) in situations associated with high level mind wandering/daydreaming and situations associated with low level of mind wandering/daydreaming | metrics are measured only one time, directly after the subject accept to participate to the study.
  demonstrate that in patients with OCD, the level of presence of obsessions is different during active and passive situations, using the THOUGHT questionnaire - scale.

SECONDARY OUTCOMES:
: Effect of OCD severity on the link between OCD and mind wandering/daydreaming | measured only one time, directly after the subject accept to participate to the study.
  Separated OCD patients in 2 groups according to their YBOCS severity to see if obsessions replace mind wandering in the same manner (the same situation and at the same level)

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Chenevier hospital, Créteil, Creteil, France